CLINICAL TRIAL: NCT00516854
Title: A Study of the Use of Combination of Anti-cholinergic and Minor Tranquilliser in the Treatment of Non-cardiac Chest Pain - a Double Blind Placebo Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC1617- 01; HARECCTR0500040
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Chest Pain
Keywords: Non-cardiac chest pain
MeSH Terms: conditions — Chest Pain | interventions — Chlordiazepoxide; clidinium

INTERVENTIONS:
Drug: chlordiazepoxide 5 mg, clidinium 2.5 mg, twice daily

SUMMARY:
Non-cardiac chest pain is a common clinical problem encountered in our practice but at present, the results of treatments are unsatisfactory. The pathogenesis remains unknown but altered motility of the esophagus and psychological factors including anxiety have been implicated as important factors. Reports of the single use of anticholinergic drugs and anxiolytics have yielded conflicting results, has been demonstrated to yield marginal or of no value. However the use of the combination therapy, especially with a double blind fashion have not been reported. On that basis, we propose to use a combination of anti-cholinergic and tranquilliser for the symptomatic treatment of non-cardiac chest pain. The aim of this study is to evaluate the efficacy of combination therapy of anti-cholinergic and anxiolytic drugs in the treatment of non-cardiac chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients over the age of 18
* Patients who are normal endoscopically
* Patients who do not have symptomatic reflux disease
* Patient who have normal coronary angiogram or patient with normal exercise radionuclide scan or patient with normal persantin radionuclide scan.

Exclusion Criteria:

* Patients with history of significant cardiac, renal, pulmonary or hepatic diseases,
* Patients with history of dyspepsia or peptic ulcer diseases
* Patient with documented reflux diseases.
* Patient on drugs that affect gastrointestinal motility in the past 2 weeks
* Patients who are pregnant or lactating
* Patients who are suffering from costochrondritis
* Patients who are known to be sensitive to benzodiazepine or anti-cholinergic
* Patients with glaucoma and benign prostatic hypertrophy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-06; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms scores, quality of life | 12 Weeks

SECONDARY OUTCOMES:
Compliance | 12 Weeks
Adverse effects | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ting Kin Cheung, Dr, Principal Investigator — Department of Medicine, Queen Mary Hospital/ The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China